CLINICAL TRIAL: NCT07029971
Title: A Phase 1a/b Clinical Trial To Determine the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Efficacy of BB-TL1A-VIAL-HLE in Healthy Adult Volunteers and in Patients With Moderate-To-Severe Ulcerative Colitis
Brief Title: A First-in-Human Study of BB-TL1A-VIAL-HLE in Healthy Adults and People With Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated based on interim analysis results indicating the primary pharmacokinetic endpoint was unlikely to be met.
Sponsor: Vial Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB-TL1A-1.0
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Phase 1a/b; Ulcerative Colitis; BB-TL1A-VIAL-HLE; Battery Bio Australia Pty Ltd
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Phase 1a: Single-ascending dose (SAD) cohorts Phase 1b: Single-arm, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A1 Cohort: 15 mg, healthy volunteers (Experimental)
  Interventions: Biological: BB-TL1A-VIAL-HLE
- A2 Cohort: 50 mg, healthy volunteers (Experimental)
  Interventions: Biological: BB-TL1A-VIAL-HLE
- A3 Cohort: 150 mg, healthy volunteers (Experimental)
  Interventions: Biological: BB-TL1A-VIAL-HLE
- A4 Cohort: 450 mg, healthy volunteers (Experimental)
  Interventions: Biological: BB-TL1A-VIAL-HLE
- B1 Cohort: TBD mg, ulcerative colitis (Active Comparator)
  Interventions: Biological: BB-TL1A-VIAL-HLE

INTERVENTIONS:
Biological: BB-TL1A-VIAL-HLE — Anti-TL1A monoclonal antibody

SUMMARY:
The goal of this clinical trial is to learn if BB-TL1A-VIAL-HLE is safe in healthy adults and is safe and effective in treating adults with moderate-to-severe ulcerative colitis. The main questions it aims to answer are:

Is the intervention safe in healthy adults and in adults with moderate-to-severe ulcerative colitis? Is the intervention effective in treating adults with moderate-to-severe ulcerative colitis? Researchers will compare the Phase 1b arm to a historical treatment arm to estimate the drug's effect size and see if the study drug is at least as effective as a relevant benchmark.

Participants will:

* Attend the clinical research site several times over the course of ~1 year
* Have blood and urine samples taken
* Undergo physical examinations
* Receive one injection of the study drug

DETAILED DESCRIPTION:
This is a Phase 1a/b integrated clinical investigation. Phase 1a is an open-label, single-ascending dose (SAD) study evaluating the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of BB-TL1A-VIAL-HLE in healthy volunteers. Phase 1b is a single-arm, open-label study evaluating the safety, PK, PD, immunogenicity, and efficacy of a single dose of BB-TL1A-VIAL-HLE in patients with moderate-to-severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria (Phase 1a)

1. Written informed consent to participate in the study and the ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures is provided.
2. Aged 18 to 55 years old (inclusive).
3. A weight of ≥50 kg and a body mass index between 18 and 32 kg/m2 (inclusive).
4. Considered healthy by the investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs.
5. Women of childbearing potential (WOCBP) may be considered if the participant is following the contraception guidance below in 5a. The participant will be questioned at each visit where there is a potential pregnancy. Similarly, male participants must follow the contraception guidance below in 5b.

   a. Female participants meet this criterion if they are: i. Postmenopausal for at least 1 year before the first dose of study drug, including a serum FSH level of >40 mIU/mL to be reported to confirm menopause.

   OR ii. Surgically sterile (documented hysterectomy [by self-disclosure] or bilateral oophorectomy ≥90 days prior to enrollment).

   OR iii. Abstinent from heterosexual intercourse as per usual lifestyle (self-reported).

   OR iv. Using effective contraceptive methods for at least 6 weeks prior to enrollment and agree to continue effective contraceptive methods throughout study participation and up to 81 weeks (t1/2 x 5) after the last dose of the study drug.

   b. Male participants meet this criterion if they agree to: i. Practice effective barrier contraception from the time of enrollment throughout study participation and up to 81 weeks (t1/2 x 5) after the last dose of the study drug.

   OR ii. Be abstinent from heterosexual intercourse as per usual lifestyle (self-reported).

   AND iii. Refrain from donating sperm during study participation and up to 81 weeks (t1/2 x 5) after the last dose of the study drug.
6. Non-smoker. If participant is a social smoker (up to 10 cigarettes per week), participant is willing to abstain during confinement.

Exclusion Criteria (Phase 1a)

1. Allergy to the investigational drug or any of its components or clinically significant allergies (excluding mild seasonal allergies), in the opinion of the investigator.
2. Use of drugs with the same target and mechanism of action as the investigational product (TL1A targeting antibodies) within 30 days or 5 half-lives (whichever is longer) prior to screening.
3. History of tuberculosis (TB) or active, latent or inadequately treated TB infection. TB testing to be conducted at screening using QuantiFERON-TB Gold. Refer to a general practitioner for X-rays, etc. if required.
4. Clinically relevant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, drug hypersensitivity, or medication history making implementation of the protocol or interpretation of the study results difficult, or that would put the participant at risk by participating in the study in the opinion of the Investigator. History or fully resolved childhood asthma with no hospitalizations, that has had no recurrence as an adult are allowed.
5. Use of prescription medications, medical devices (other than hormonal contraception [e.g., oral contraceptive pills, long-acting implantable hormones, or injectable hormones], vaginal ring, or IUD) within 30 days prior to enrollment, or use of any over-the-counter (OTC) medications, herbal remedies, supplements, or vitamins within 30 days prior to enrollment and during the course of the study without prior approval of the Investigator and the independent Medical Monitor. Use of simple analgesics (e.g., paracetamol, a nonsteroidal anti-inflammatory drug [NSAID]) and antihistamines may be permitted at the discretion of the Investigator.
6. Evidence of malignancy or other clinically relevant abnormality in the opinion of the investigator at screening or within 5 years prior to Day 1, with the exception of squamous cell or basal cell carcinomas.
7. Known or suspected autoimmune disorder.
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCV Ab).
9. Administered a live attenuated vaccine within 28 days of enrollment (participants must also abstain from taking any live vaccines until at least 12 weeks after study completion).
10. A hospital admission or major surgery within 30 days prior to screening.
11. Participation in any other investigational drug trial within 30 days prior to screening or 5 half-lives, whichever is longer.
12. Confirmed or suspected COVID-19 infection within 14 days of any screening procedures.
13. Substance use disorder (SUD) and/or alcohol use disorder (AUD).
14. Other conditions that may affect compliance in the opinion of the investigator, or who is unable to participate in the study on his/her own.
15. The possible sites of injection (abdomen, front of thighs) have tattoos, scars, or significant dermatological disorders that prohibit the clear assessment of injection site reactions.
16. Blood donation ≤30 days prior to screening.
17. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN) at baseline.
18. Serum total bilirubin >2 times ULN at baseline.
19. Neutrophil count below 1,000 cells/µL at baseline.
20. Urea or serum creatinine >1.5 times ULN at baseline.
21. Employees or related personnel of the investigator, study site, or sponsor.

Inclusion Criteria (Phase 1b)

1. Written informed consent to participate in the study and the ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures is provided.
2. Age ≥ 18 years.
3. A weight ≥ 50 kg and a body mass index (BMI) between 18 and 32 kg/m2 (inclusive).
4. Women of childbearing potential (WOCBP) and men must follow the contraception guidance as per the original protocol, ensuring no potential for pregnancy.
5. A confirmed diagnosis of UC for ≥ 3 months.
6. Moderate-to-severe UC, as defined by:

   1. Aggregate UC severity score ≥ 4
   2. Endoscopic severity score ≥ 2
   3. Blood in stool score ≥ 1
7. Active disease beyond the rectum, with > 15 cm of active disease from the anal verge (confirmed by endoscopy).
8. Documented inadequate response, loss of response, or intolerance to ≥ 1 prior therapy from any of the following classes, confirmed by medical record OR investigator attestation OR patient-reported history (Investigator must confirm in the eCRF):

   1. Systemic corticosteroids
   2. Immunosuppressants
   3. Anti-TNF agents
   4. Anti-integrin inhibitors
   5. Anti-IL-12/23 inhibitors
   6. JAK inhibitors
   7. S1PR modulators
9. If concomitantly taking 5-aminosalicylates, the participant must be on a stable dose for at least 4 weeks before baseline efficacy assessments.*
10. If concomitantly taking low-dose corticosteroids (≤ 20 mg/day), the participant must be on a stable dose for at least 2 weeks before baseline efficacy assessments.*
11. If concomitantly taking thiopurines, the participant must be on a stable dose for at least 8 weeks before baseline efficacy assessments.* *Baseline efficacy assessments include 7-Day Symptom Collection and Endoscopy.

Exclusion Criteria (Phase 1b)

1. Diagnosis of Crohn's disease, indeterminate colitis, or UC limited to the rectum (< 15 cm from the anal verge).
2. Current evidence of fulminant colitis, toxic megacolon, or bowel perforation.
3. Active, serious infection requiring IV antibiotics within 4 weeks prior to enrollment.
4. History of cancer within 5 years, except for:

   1. Cured non-melanoma skin cancer, OR
   2. Localized cervical cancer treated definitively.
5. Hemaglobin < 8.0 g/dL at baseline.
6. Neutrophil count < 1.0 x 109/L at baseline.
7. Platelet count < 100 x 109/L at baseline.
8. Serum creatinine > 2x ULN at baseline.
9. ALT or AST > 3x ULN at baseline.
10. Total bilirubin > 2x ULN at baseline, unless the participant has a documented history of Gilbert's syndrome.
11. History of clinically significant drug or food allergy, including anaphylaxis or serious adverse reactions (excluding mild seasonal allergies).
12. History of untreated or inadequately treated latent or active tuberculosis (TB), or a positive QuantiFERON-TB Gold test at screening without prior appropriate therapy.
13. Positive test for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), or hepatitis C antibody (anti-HCV) at screening.
14. Receipt of a live attenuated vaccine within 28 days prior to the first dose of investigational product.
15. History of alcohol use disorder or substance use disorder (excluding nicotine or caffeine) within the past 12 months, as defined by DSM-5 criteria, that may interfere with study participation or pose additional risk.
16. Major surgery or hospitalization for any reason (excluding UC-related procedures) within 30 days prior to screening.
17. Use of investigational drugs or devices within 30 days of baseline efficacy assessments or 5 half-lives, whichever is longer.*
18. Use of biologics within 12 weeks of baseline efficacy assessments or 5 half-lives, whichever is longer.*
19. Use of rituximab within 1 year of baseline efficacy assessments.*
20. Use of parenteral corticosteroids within 4 weeks or rectal administration of corticosteroids within 2 weeks of baseline efficacy assessments.*
21. Rectal administration of 5-aminosalicylates within 2 weeks of baseline efficacy assessments.*
22. Use of tacrolimus, methotrexate, cyclosporine, mycophenolate mofetil, immunoadsorption columns, d-penicillamine, leflunomide, thalidomide, fish-oil preparations, probiotics, fecal transplantation, nonsteroidal anti-inflammatory agents (NSAIDs), and/or aspirin > 31 mg/day within 2 weeks of baseline efficacy assessments.*
23. Employees or related personnel of the investigator, study site, or sponsor. *Baseline efficacy assessments include 7-Day Symptom Collection and Endoscopy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting or intolerable treatment related adverse events | From enrollment to the end of the follow up period at Day 355
Incidence, severity and causal relationship of treatment emergent AEs (TEAEs) and withdrawals due to TEAEs | From enrollment to the end of the follow up period at Day 355
Incidence and magnitude of abnormal laboratory findings | From enrollment to the end of the follow up period at Day 355
Abnormal and clinically relevant changes in vital signs, blood pressure and electrocardiogram parameters | From enrollment to the end of the follow up period at Day 355
Percentage of participants who achieve endoscopic improvement at 12 weeks post-dose (Ph-1b) | From enrollment to end of induction period at 12 weeks
  (defined as an endoscopic severity score* of ≤1 with no friability)
  *The endoscopic severity score range is 0-3 with a higher score indicating higher severity.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | From enrollment to end of follow up period at Day 355
Time at which maximum plasma concentration is observed (Tmax) | Enrollment to end of follow up period at Day 355
Area under the plasma concentration-time profile from time zero to Day 15 (AUCDay15) | Enrollment to end of follow up period on Day 355
Area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (AUClast) | Enrollment to end of follow up period at Day 355
Area under the plasma concentration-time curve extrapolated to infinity (AUCinf) | Enrollment to end of follow up period at Day 355
Dose normalized maximum plasma concentration (Cmax[dn]) | Enrollment to end of follow up period at Day 355
Dose normalized area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (AUClast[dn]) | Enrollment to end of follow up period at Day 355
Half-life (t½) | Enrollment to end of follow up period at Day 355
Mean residence time (MRT) | Enrollment to end of follow up period at Day 355
Systemic clearance (CL) | Enrollment to end of follow up period at Day 355
Volume of distribution at steady state (Vss) | Enrollment to end of follow up period at Day 355
Percentage of participants who achieve clinical remission at 12 weeks post-dose (Ph-1b) | Baseline to 12 weeks post-dose
  (defined as an endoscopic severity score* of ≤ 1, ≥ 1-point decrease from baseline to achieve a bowel movement frequency score** of ≤ 1, and blood in stool score*** of 0)
  *The endoscopic severity score range is 0-3 with a higher score indicating higher severity.
  **The bowel movement frequency score range is 0-3 with a higher score indicating higher severity.
  ***The blood in stool score range is 0-3 with a higher score indicating higher severity.
Percentage of participants who achieve clinical response at 12 weeks post-dose (Ph-1b) | Baseline to 12 weeks post-dose
  (defined as a decrease from baseline in the aggregate ulcerative colitis severity score* of ≥ 2 points and ≥30% reduction from baseline, and a decrease in blood in stool score** of ≥ 1 or an absolute blood in stool score of ≤ 1)
  *The aggregate ulcerative colitis severity score range is 0-9 comprised of three subscores (blood in stool score, bowel movement frequency score, and endoscopic severity score) with a higher score indicating higher severity of ulcerative colitis.
  **The blood in stool score range is 0-3 with a higher score indicating higher severity.
Percentage of participants who achieve symptomatic remission at 12 weeks post-dose (Ph-1b) | Baseline to 12 weeks post-dose
  (defined as a bowel movement frequency score* of 0 and blood in stool score** of 0)
  *The bowel movement frequency score range is 0-3 with a higher score indicating higher severity.
  **The blood in stool score range is 0-3 with a higher score indicating higher severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Dymocks Building, WellShare Site, Sydney, New South Wales
  - Arcadia Pittwater Private Hospital (Operated by Battery Bio), Warriewood, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided